CLINICAL TRIAL: NCT03984058
Title: Comparing Recruitment Strategies for a Randomized Controlled Trial in Sleep Apnea and Prediabetes
Brief Title: Recruitment Strategies Comparing Different Strategies in Sleep Apnea and Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Fusion Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00199862
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2020-11

CONDITIONS: Sleep Disorder; Pre Diabetes; Obstructive Sleep Apnea
Keywords: Pre-diabetes; Sleep Apnea; PAP Therapy; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Wake Disorders; Glucose Intolerance; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Arm 1 (Other): All enrolled participants will have participants' PAP usage monitored by Fusion Health using the ResMed AirView Remote Monitoring system. Fusion Health will provide individual care for each participant by monitoring daily PAP usage by all study participants. This assessment ensures routine follow-up of PAP adherence during the study. The responsibility for patient care during the study, however, will fall on clinical site staff with any needed assistance by the Fusion Health staff. An intervention will be required when PAP adherence decreases or if any other issues are identified that require a face-to-face visit.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — A lifestyle intervention program adapted from the Diabetes Prevention Program (DPP). Study participants will start lifestyle intervention on the day of initiating PAP therapy. The 3-month program will be followed: Patient-facing Online Platform: The program will be accessible to study participant via the Web or a Web application available for the Android and iOS devices. Behavioral Weight Loss Goals and Lessons: The program begins with an introductory session that presents the basic goals for the program followed by 12 weekly multimedia lessons. Submission of self-monitoring data: Participants will submit daily weight, caloric intake, and physical activity minutes at least weekly to the study website for 12 weeks. Automated Feedback: In response to the self-monitoring data, participants receive a weekly automated message that compares participants' self-reported values to participants' goals for weekly and overall weight loss, caloric intake, and physical activity minutes.

SUMMARY:
Recruitment strategies comparing different strategies.

DETAILED DESCRIPTION:
Patients with prediabetes and moderate-to-severe Obstructive Sleep Apnea (OSA). To determine the recruitment yields from electronic medical record (EMR) vs the general community. To assess the adherence to positive airway pressure (PAP) therapy among patients with prediabetes and moderate-to-severe OSA.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetes: A1c value of 6.0-6.4% and fasting glucose of 100-125 mg/dl
* Moderate-to-severe OSA [4% oxygen desaturation index (ODI) ≥ 20/h]
* Ability to provide informed consent
* Able to comply with all study procedures and be available for the study duration
* Availability of smart phone

Exclusion Criteria:

* BMI < 28 or ≥ 38 kg/m2
* Type 1 or Type 2 diabetes mellitus
* Pregnancy
* Use of glucose-lowering or weight loss medications (e.g., metformin, orlistat, phentermine)
* Prior or anticipated bariatric surgery
* Current use of PAP or oral appliance therapy for OSA
* Commercial driver
* Report of a motor vehicle accident or near-miss due to sleepiness within 2 years
* Epworth Sleepiness Scale score10 > 18
* Current (prevalent) use of oral corticosteroids (within 1 month)
* Participation in a concurrent clinical trial
* Unstable medical conditions: uncontrolled angina and/or congestive heart failure, uncontrolled blood pressure or resistant hypertension [BP ≥ 160/100 among those with hypertension, requiring 3 or more meds], severe chronic obstructive pulmonary disease, cancer, or active psychiatric disease
* Other sleep disorders (e.g., circadian rhythm disorder, working night or rotation shift, short sleep duration based on self-reported habitual sleep patterns < 5 hrs/night)
* Use of supplemental oxygen during wakefulness or sleep
* Central sleep apnea (central apnea index ≥ 5/h) or Cheyne-Stokes respiration (> 10 minutes of continues period breathing) on the screening home sleep test Resting awake SpO2 < 90%
* Chronic opiate use.
* Use of illicit drug / marijuana use more than once per week
* Difficulty understanding or speaking English
* Anything that, in the opinion of the site investigator, would place the participant at increased risk or preclude a participant's ability to adhere to study protocols or complete the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Recruitment Yield as assessed by number of participants enrolled from electronic medical records (EMR) | 1 year
  Determine recruitment yield from EMR versus the general community.

SECONDARY OUTCOMES:
Adherence to Pap Therapy as assessed by the ResMed AirView Remote Monitoring system | 1 Week
  Participants will have PAP usage monitored with the ResMed AirView Remote Monitoring system. An intervention will be required when PAP adherence decreases or if any other issues are identified that require a face-to-face visit. A phone contact or in-person visit will be scheduled if the following findings observed for ≥3 consecutive nights:
  * Suboptimal adherence (< 5 hours per night);
  * Mean leak is high (> 20 L/min); or treatment is not optimal (AHI ≥ 5 events/h)
  Each participant will have a follow-up visit ~ 7 days after starting PAP therapy

CONTACTS AND LOCATIONS:
Overall Officials: Naresh Punjabi, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Department of Medicine, Johns Hopkins University, Baltimore, Maryland, United States